CLINICAL TRIAL: NCT01614002
Title: Open, Multicenter Observational Study of Docetaxel Utilized in Mono- or Combination Therapy for Treatment of Breast Cancer, NSCLC, Prostate Carcinoma, Adenocarcinoma of Stomach and Advanced Squamous Cell Carcinoma of Head/Neck Region.
Brief Title: A Non Interventional Study With Doce Onkovis (Docetaxel) Utilized for the Treatment of Cancer
Status: Completed | Type: Observational
Sponsor: Onkovis GmbH (Industry)
Collaborators: AKP Freiburg GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ONKODOC 01
Record Dates: First submitted 2012-06-01; First posted 2012-06-07 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Carcinoma
Keywords: carcinoma; breast cancer; non-small cell lung cancer; prostata cancer; adenocarcinoma of the stomach; squamous cell carcinoma of the head and neck region; ambulant chemotherapy; treatment cycles; Docetaxel; Doce onkovis; Quantity of Docetaxel; Packaging Sizes
MeSH Terms: conditions — Carcinoma; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- carcinoma, Doce onkovis (Docetaxel): treatment in mono- or combination therapy with Docetaxel of breast cancer, non-small cell lung cancer, prostata carcinoma, adenocarcinoma of the stomach and advanced squamous cell carcinoma of the head/neck region.

SUMMARY:
The main purpose of this observational study with Docetaxel is to determine the number of treatment cycles and the quantity of Doce onkovis needed therefore under the special circumstance of ambulant chemotherapy.

onkovis aims an economical utilization of the chemotherapeutics.The provision with adapted packaging sizes as to decrease the excess quantity to be discarded follows also this objective.

Secondary objectives are the evaluation of the safety and tolerability of Doce onkovis. To this purpose data regarding co medications and adverse events are also collected.

ELIGIBILITY:
Inclusion Criteria:

* Indication for Docetaxel according to the SmPC and treating physician

Exclusion Criteria:

* according to the Docetaxel SmPC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated in practices, clinics, hospitals
Sampling Method: Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
the quantity of Doce onkovis needed pro treatment cycle | the time the participants will be followed depends on the number of treatment cycles; that means the time frame may extend up to 24 weeks (8 cycles).
  Determine the quantity of Doce onkovis needed pro treatment cycle

SECONDARY OUTCOMES:
adverse events during and after treatment | up to 24 weeks (8 cycles)
  The number and kind of adverse events during and after the intra-venous application of Docetaxel will be assessed and documented.

CONTACTS AND LOCATIONS:
Locations (23):
- Germany (23):
  - Practice, Berlin
  - Practice, Brandenburg
  - Practice, Chemnitz
  - Practice, Cottbus
  - Practice, Dresden
  - Practice, Elstra
  - Practice, Freital
  - Practice, Fürstenwalde
  - Practice, Halle
  - Practice, Köthen
  - Practice, Kronach
  - Hospital, Leipzig
  - Practice, Leipzig
  - Practice, Magdeburg
  - Practice, Meiningen
  - Practice, Mühlhausen
  - Practice, Parchim
  - Practice, Plauen
  - Practice, Scheibenberg
  - Clinic, Torgau
  - Practice, Werdau
  - Practice, Zittau
  - Practice, Zwickau